# Study Title for Study Participants: Testing perfusion CT to predict response to bevacizumab treatment for ovarian, fallopian tube and peritoneal cancers

Official Study Title for Internet Search on <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>: EAE161 Perfusion CT to Predict Progression-free Survival and Response Rate in Bevacizumab and Paclitaxel Treatment of Platinum-Resistant Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Carcinoma.

#### **Screening Consent**

Version Date: June 13, 2018

# What is the usual approach to monitoring my ovarian, fallopian tube or peritoneal carcinoma cancer?

You are being asked to take part in this research study because you are about to receive a CT exam of your chest, abdomen and pelvis as part of your routine care. The exams are being obtained to see whether your ovarian, fallopian tube or peritoneal cancer can be seen with imaging. If the CT exam indicates that you have persistent or recurrent cancer, your doctor would like to send the CT images and information on your tumor type to researchers at the ECOG-ACRIN Cancer Research Group, a National Cancer Institute research group. The ECOG-ACRIN scientists will look at your CT images to see if you are eligible to participate in an ECOG-ACRIN imaging study. If you are found to be eligible, your doctor will explain to you the imaging study and, if you choose to participate at that time, you will be asked to agree to a separate consent.

### What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices for your care. For example:

- you may choose to have the usual routine care
- you may choose to take part in a different research study, if one is available

### Why is this study being done?

The purpose of this is to obtain your permission to screen you for eligibility to a trial. We are asking permission to submit images from your chest abdomen and pelvic CT exam to ECOG-ACRIN. These images will be looked at to see whether you are eligible for an imaging trial

testing perfusion CT. Perfusion CT is an imaging test that looks at the blood flow to your tumor. Contrast agent is injected into your veins while you are in the scanner and many sequential images of your tumor are obtained while the contrast flows into then out of your tumor. The experience for you is similar to the conventional CT exam except the images taken for this study are more focused in a specific area of your body, where the tumor is located.

If this screening finds that you are eligible, the imaging study will be explained to you separately. At that time, if you choose to participate in the imaging study, you will be asked to sign another consent. If you are not found to be eligible on screening, you will no longer be in this study. You will be treated with the usual routine care.

There will be about 300 patients who will be screened.

#### What are the study groups?

All participants in the screening study will receive a CT scan as part of the usual care. If you have recurrent or persistent cancer on your CT scan, your scan will be used to see if you have a lesion that makes you eligible for an imaging study to test perfusion CT. These CT images will be submitted to ECOG-ACRIN where it will be confirmed if you are eligible for the ECOG-ACRIN imaging study.

Another way to find out what will happen to you during this research study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.

#### **Screening**



### How long will I be in this study?

Once your images from your CT scan have been sent to ECOG-ACRIN, the scan will be reviewed by ECOG-ACRIN within five business days. ECOG-ACRIN will then let your

doctor know if you are eligible for the perfusion CT imaging study. If eligible, a separate discussion and consent process will take place. If you are found eligible and are enrolled in the study, participation in that study would be a minimum of 18 months and a maximum of three and a half years.

#### What extra tests and procedures will I have if I take part in this study?

You will need a blood test to look at your kidney function. The scan you are receiving is part of usual care for your cancer.

#### What possible risks can I expect from taking part in this study?

If you choose to take part in this research study, there is a risk that:

- Disclosure and misuse of your health information. This is a small risk as your health information is protected, but there is always a risk.
- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- If your CT scan shows tumor, your treatment may be delayed by up to five days while awaiting results from this screening.

#### What possible benefits can I expect from taking part in this study?

This screening is not expected to be of benefit to you.

## Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB or FDA.

## What are my rights in this study?

Taking part in this research study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care

#### What are the costs of taking part in this study?

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this research study, including the cost of study drug preparation and administration, tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are being done at no charge. Before you decide to be in the research study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this screening research study. The review of your CT scan at ECOG-ACRIN will be completed at no cost to you or your insurance. You will not be responsible for the cost of the CT perfusion exam, the kidney function and the CA125 blood tests.

#### What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this research study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for research study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a research study.

## Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

The ECOG-ACRIN Cancer Research Group is conducting this study. ECOG-ACRIN is a cancer research group that conducts studies for the National Cancer Institute. Your doctor is a member of ECOG-ACRIN or another group that is participating in this study. To help protect your privacy, ECOG-ACRIN has obtained a Confidentiality Certificate from the Department of Health and Human Services (DHHS). With this Certificate, ECOG-ACRIN

cannot be forced (for example, by court subpoena) to disclose information that may identify you in any federal, state or local civil, criminal, administrative, legislative or other proceeding. Disclosure will be necessary, however, upon request of DHHS for audit or program evaluation purposes.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.
- Harvard Tumor Metrics Imaging Core
- ECOG-ACRIN Cancer Research Group

#### Where can I get more information?

You may visit the NCI Web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### Who can answer my questions about this study

| You can talk to the study doctor a | about any questions or concerns you | have about this study o |
|---|---|---|
| to report side effects or injuries. ( | Contact the study doctor | (insert name |
| of study doctor[s]) at | (insert telephone number). | |
| My signature agreeing to take | part in the study | |
| | and it read to me. I have discussed it wered. I will be given a signed copy of this study. | • |
| Participant's signature | | |
| Date of signature | | |

| Signature of person(s) conducting the informed consent discussion |
|-------------------------------------------------------------------|
| Date of signature |

# Study Title for Study Participants: Testing perfusion CT to predict response to bevacizumab treatment for ovarian, fallopian tube and peritoneal cancers

Official Study Title for Internet Search on <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>: EAE161 Perfusion CT to Predict Progression-free Survival and Response Rate in Bevacizumab and Paclitaxel Treatment of Platinum-Resistant Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Carcinoma.

#### **Imaging Consent**

Version Date: June 13, 2018

# What is the usual approach to monitoring my treatment for ovarian, fallopian tube or peritoneal carcinoma cancer?

You are being asked to take part in this research study because you have recurrent or persistent epithelial ovarian, tubal or peritoneal cancer. Your physician is considering treating you with paclitaxel and bevacizumab and one of your lesions has been found eligible to receive perfusion CT. Researchers at the ECOG-ACRIN Cancer Research Group, part of the National Cancer Institute's research groups, want to find out if perfusion CT imaging can predict how well your cancer responds to paclitaxel and bevacizumab treatment.

### What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices for your care. For example:

- you may choose to have the usual routine care
- you may choose to take part in a different research study, if one is available

### Why is this study being done?

The purpose of this research study is to study perfusion CT and how it works in combination with your disease and treatment. Perfusion CT imaging looks at the blood flow to your tumor. Contrast agent is injected into your veins while you are in the scanner and many sequential images of your tumor are obtained while the contrast flows in and out of your tumor.

The experience for you in the scanner is similar to the conventional CT exam except imaging will take a bit longer (e.g. ~20-30 minutes). The exam will be performed in two parts and the

contrast injected will also be administered through a vein at two different time points. We will first focus on imaging a specific tumor nodule several times while the contrast is flowing in and out of it; then, after a 10 minute wait, a second administration of contrast will be given and one set of images of your torso will be obtained. The total amount you receive with the two administrations will be similar to that for a conventional CT exam.

If this study shows that CT perfusion results are related to the effectiveness of the tumor treatment, investigators will be able to use perfusion CT exams in the future to predict whether a certain drug is likely be successful in a patient with ovarian, fallopian tube or primary peritoneal cancer early on in the course of therapy. There will be about 184 people who will receive CT perfusion as part of this research study.

#### What are the study groups?

All participants will receive the same study intervention. You will have a perfusion CT scan prior to receiving bevacizumab and another perfusion CT scan after starting bevacizumab. Another way to find out what will happen to you during this research study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.



## Rev Add! How long will I be in this study?

You will receive your first perfusion CT within 7 days before you start your chemotherapy treatment. A second perfusion CT will be performed within 17 days after starting bevacizumab + paclitaxel and before your second dose of bevacizumab. You will be followed through the course of your chemotherapy treatment and receive routine imaging every 9 weeks the first year you are on this study. After that you will receive routine standard of care imaging every 12 weeks while on study. Your doctor will continue to follow you for up to 18 months after the last patient is enrolled on this study or you withdraw consent. Your follow-up may be completed in various ways; during imaging sessions, clinic visits and/or phone calls. You will be on this study for a minimum of 18 months to a maximum three and a half years. For the first two years you will be followed every three months. After two years, follow-up will go to every six months.

## What extra tests and procedures will I have if I take part in this study?

Most of the exams, tests, and procedures you will have are part of the usual care for your cancer. However, there are some extra tests that you will receive as part in this research study.

#### **During the study:**

If you choose to take part in this study, then you will need the following extra test and procedures. They are not part of the usual care for your type of cancer.

These extra tests include:

- Perfusion CT for a total of two exams
- Blood tests of your CA-125 level twice (within 2 days <u>before or after each</u> perfusion scan). CA-125 is to measure the amount of CA-125 protein in your blood.

### What possible risks can I expect from taking part in this study?

If you choose to take part in this research study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- Your treatment may be delayed by up to five days for the imaging portion of this study.
- The iodinated contrast you receive as part of the perfusion CT may affect how different parts of your body work such as your kidneys.

The perfusion CT that you will receive in this study will expose you to extra radiation that is equal to about 4 years' worth of background radiation. The radiation dose from a perfusion CT exam is similar in amount to that of a standard CT exam that your doctor uses to measure your tumor. However, as we are scanning only a specific portion of your body, the radiation dose to that area may be up to two times higher. In total, the added radiation from the two perfusion CT exams of this study will be about the same as three added standard CT exams, but will be administered to a specific portion of your body For medical imaging exams, you are exposed to low levels of radiation. It is not known for certain what the health risk of this radiation is. However, it is expected that the risk of potentially getting a new cancer due the radiation doses used here for diagnostic imaging is less than 1:1,000, and is likely much lower.

Perfusion CT does require that we place an intravenous (IV) catheter and give a contrast agent (also called X-ray dye). In this study you will be given contrast and that is split into two administrations during the perfusion CT exam. The total amount of contrast given is the same as for a standard CT. The tables below shows the most common and the most serious side effects that researchers know about that might occur with this:

#### Risks Associated With Intravenous (IV) Catheter Placement

#### **COMMON**

In 100 people receiving an IV needle placement to give contrast agent, more than 20 and up to 100 may have:

- Minor discomfort
- Bruising
- Pain at the injection site
- Leaking of contrast agent from IV needle

#### RARE, MAY BE SERIOUS

In 100 people receiving an IV needle placement to give contrast agent, 1 or fewer may have:

- Fainting
- Bleeding

#### Risks Associated with the Contrast Agent or X-Ray Dye

#### OCCASIONAL, MAY BE SERIOUS

In 100 people receiving contrast agent or x-ray dye, 4 to 20 people may have:

- Nausea/vomiting;
- Warm sensation or a flushed feeling;
- Skin rashes or hives
- Itching

#### RARE, MAY BE SERIOUS

In 1,000 people receiving contract agent or x-ray dye, 1 or fewer may have:

• Temporary damage to the kidney

#### **VERY RARE AND SERIOUS**

In 1,000,000 people receiving contract agent or x-ray dye, 4 or fewer may have:

- Swelling of the mouth and throat
- Abnormal heart rhythm
- Fainting and very low blood pressure requiring treatment

There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

#### What possible benefits can I expect from taking part in this study?

This research study has only a small chance of helping you because we do not know if the perfusion CT exam accurately predicts the effects of the bevacizumab drug. This research study may help researchers learn things that may help other people in the future.

#### Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB or FDA.

### What are my rights in this study?

Taking part in this research study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

| For questions about your rights while in this study, call the | |
|---|---|
| (insert name of center) Institutional Review Board at | (insert telephone |
| <mark>number)</mark> . (Note to Local Investigator: Contact information for patient rep | resentatives or |
| other individuals at a local institution who are not on the IRB or research | team but take calls |
| regarding clinical trial questions can also be listed here.) | |

### What are the costs of taking part in this study?

You will not be charged for the two perfusion CT exams while you take part in this research study.

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this research study, including the cost of study drug preparation and administration, tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are being done at no charge. Before you decide to be in the research study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this research study.

#### What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this research study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for research study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a research study.

#### Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

The ECOG-ACRIN Cancer Research Group is conducting this study. ECOG-ACRIN is a cancer research group that conducts studies for the National Cancer Institute. Your doctor is a member of ECOG-ACRIN or another group that is participating in this study. To help protect your privacy, ECOG-ACRIN has obtained a Confidentiality Certificate from the Department of Health and Human Services (DHHS). With this Certificate, ECOG-ACRIN cannot be forced (for example, by court subpoena) to disclose information that may identify you in any federal, state or local civil, criminal, administrative, legislative or other proceeding. Disclosure will be necessary, however, upon request of DHHS for audit or program evaluation purposes.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- ECOG-ACRIN Cancer Research Group
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.
- Harvard Tumor Imaging Metrics Core

### Where can I get more information?

You may visit the NCI Web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>, as required

by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| bout this study? | |
|---|---|
| ut any questions or concerns y tact the study doctor | (insert name |
| (insert telephone nun | <mark>nber)</mark> . |
| art in the main study | |
| it read to me. I have discussed d. I will be given a signed co | • |
| e informed consent discussion | n |
| 1 1 i | at any questions or concerns that the study doctor (insert telephone number tin the main study) It read to me. I have discussed. I will be given a signed content of the study of the stu |

# Título del estudio para los participantes del estudio: Evaluación de la TAC de perfusión para predecir la respuesta al tratamiento con bevacizumab en cáncer de ovarios, de trompas de Falopio y peritoneal

## Título oficial del estudio para la búsqueda en Internet en

https://ClinicalTrials.gov: EAE161 Perfusion CT to Predict Progression-free Survival and Response Rate in Bevacizumab and Paclitaxel Treatment of Platinum-Resistant Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Carcinoma.

(EAE161 TAC de perfusión para predecir la supervivencia libre de progresión y la tasa de respuesta al tratamiento con bevacizumab y paclitaxel en carcinoma ovárico epitelial, de trompas de Falopio o peritoneal resistente a platino persistentes o recurrentes).

#### Consentimiento para la realización de pruebas de diagnóstico por imágenes

Fecha de la versión: 13 de junio de 2018

# ¿Cuál es el enfoque habitual para el monitoreo del tratamiento del cáncer ovárico, de trompas de Falopio o peritoneal?

Se la invita a participar en este estudio de investigación porque tiene cáncer ovárico epitelial, en las trompas de Falopio o peritoneal recurrente o persistente. Su médico está considerando tratarla con paclitaxel y bevacizumab y se ha determinado que una de las lesiones es apta para recibir una tomografía computada (TAC) de perfusión. Los investigadores del grupo ECOG-ACRIN Cancer Research Group, parte de los grupos de investigación del Instituto Nacional del Cáncer, desean averiguar si la evaluación mediante TAC de perfusión puede predecir qué tan bien responde su cáncer al tratamiento con paclitaxel y bevacizumab.

### ¿Cuáles son mis otras opciones si no participo en este estudio?

Si decide no participar en este estudio, tiene otras opciones para su atención. Por ejemplo:

- puede optar por recibir la atención habitual de rutina
- puede optar por participar en un estudio de investigación diferente, si hubiera uno disponible

#### ¿Por qué se realiza este estudio?

El objetivo de este estudio de investigación es evaluar la TAC de perfusión y la forma en que esta funciona en combinación con su enfermedad y tratamiento. La TAC de perfusión observa el flujo de sangre al tumor. Mientras está en el equipo de tomografía, se le inyecta un agente de contraste en las venas y se obtienen muchas imágenes secuenciales de su tumor mientras el contraste fluye dentro y fuera del tumor.

Para usted, la experiencia dentro del equipo será similar a un examen de TAC convencional, salvo que tomará un poco más de tiempo (p. ej., ~20-30 minutos). El examen se dividirá en dos partes y el contraste que se inyecte también se administrará por medio de una vena en dos momentos diferentes. Inicialmente, nos concentraremos en obtener imágenes de un nódulo tumoral específico varias veces mientras el contraste fluye dentro y fuera del tumor; después, tras una espera de 10 minutos, se realizará una segunda administración de contraste y se obtendrá un conjunto de imágenes del torso. La cantidad total que reciba con las dos administraciones será similar a la de una tomografía convencional.

Si este estudio demuestra que los resultados de la TAC de perfusión están relacionados con la efectividad del tratamiento del tumor, en el futuro, los investigadores podrán utilizar exámenes de TAC de perfusión para predecir si un fármaco determinado podría funcionar en un paciente con cáncer ovárico, de trompas de Falopio o peritoneal primario en las etapas iniciales del tratamiento. Como parte de este estudio de investigación, aproximadamente 184 personas recibirán TAC de perfusión.

#### ¿Cuáles son los grupos del estudio?

Todos los participantes recibirán la misma intervención del estudio. Se le realizará una TAC de perfusión antes de que reciba bevacizumab y otra TAC de perfusión después del inicio de bevacizumab. Lea el cuadro a continuación como otra manera de conocer qué le pasará durante este estudio de investigación. Empiece a leer de izquierda a derecha, siguiendo las líneas y flechas.



Rev. Add1

# ¿Durante cuánto tiempo participaré en este estudio?

Se le realizará su primera TAC de perfusión dentro de los 7 días previos al inicio de su tratamiento con quimioterapia. La segunda TAC de perfusión se le realizará dentro de los 17 días después del inicio del tratamiento con bevacizumab + paclitaxel y antes de la segunda dosis de bevacizumab. Se le realizará seguimiento durante su tratamiento de quimioterapia y estudios de diagnóstico por imágenes de rutina cada 9 semanas durante el primer año que participe en este estudio. Después de eso, se le realizarán estudios de diagnóstico por

imágenes convencionales de rutina cada 12 semanas mientras participe en el estudio. Su médico seguirá realizándole seguimiento por hasta 18 meses después de la inscripción del último paciente en este estudio o hasta que usted retire su consentimiento. El seguimiento podrá realizarse de diferentes maneras: durante las sesiones en que se realicen estudios de diagnóstico por imágenes, en visitas a la clínica o a través de llamadas telefónicas. Participará en este estudio por un mínimo de 18 meses hasta un máximo de tres años y medio. Durante los primeros dos años, se le realizará seguimiento cada tres meses. Después de dos años, el seguimiento se hará cada seis meses.

# ¿Qué pruebas y procedimientos adicionales se me realizarán si participo en este estudio?

La mayoría de los exámenes, las pruebas y los procedimientos que se le harán forman parte de la atención habitual para su cáncer. Sin embargo, como parte de este estudio de investigación, se le realizarán algunas pruebas adicionales.

#### **Durante el estudio:**

Si decide participar en este estudio, tendrá que realizarse las siguientes pruebas y procedimientos adicionales. Estos no forman parte de la atención habitual para su tipo de cáncer.

Estas pruebas adicionales incluyen las siguientes:

- Dos TAC de perfusión
- Análisis de sangre para detectar sus niveles de CA-125 dos veces (dentro de los 2 días antes o después de cada TAC de perfusión). Este análisis mide la cantidad de proteína CA-125 en la sangre.

# ¿Cuáles son los posibles riesgos que puedo esperar de la participación en este estudio?

Si decide participar en este estudio de investigación, existe el riesgo de lo siguiente:

- Pueda perder tiempo de trabajo o en su hogar y pasar más tiempo en el hospital o en el consultorio médico de lo habitual
- El tratamiento puede demorarse hasta cinco días para que pueda realizarse la porción de obtención de imágenes de este estudio.
- El contraste yodado que se le administre como parte de la TAC de perfusión puede afectar el funcionamiento de distintas partes del cuerpo, por ejemplo, los riñones.

La TAC de perfusión que recibirá en este estudio la expondrá a una radiación adicional que equivale a, aproximadamente, 4 años de radiación ambiental. La dosis de radiación de una TAC de perfusión es similar a la cantidad que recibe en una TAC estándar utilizada por su médico para medir el tumor. Sin embargo, dado que estamos analizando solo una porción específica de su cuerpo, la dosis de radiación de esa área puede ser hasta dos veces más alta. En total, la radiación adicional de las dos TAC de perfusión de este estudio será casi la

misma que tres TAC estándares sumadas, pero se administrará en una porción específica del cuerpo. En el caso de los exámenes médicos de diagnóstico por imágenes, usted queda expuesta a bajos niveles de radiación. No se conoce con certeza cuál es el riesgo de esta radiación para la salud. Sin embargo, se espera que el riesgo potencial de contraer un nuevo cáncer debido a las dosis de radiación utilizadas aquí para las pruebas de diagnóstico por imágenes es inferior a 1:1000 y, posiblemente, sea mucho más bajo.

La TAC de perfusión requiere la colocación de un catéter intravenoso (IV) y la administración de un agente de contraste (también llamado tinte radiográfico). En este estudio, durante la TAC de perfusión, se le administrará contraste dividido en dos dosis. La cantidad total de contraste administrado será la misma que para una TAC estándar. Las siguientes tablas muestran los efectos secundarios más frecuentes y más graves que los investigadores conocen sobre lo que podría ocurrir con:

#### Riesgos asociados a la colocación del catéter intravenoso (IV)

#### **FRECUENTES**

En 100 personas a quienes se les ha colocado una aguja intravenosa para la administración de un agente de contraste, más de 20 y hasta 100 personas pueden tener:

- Molestias menores
- Hematomas
- Dolor en el lugar de la inyección
- Drenaje (goteo) del agente de contraste desde la aguja IV

#### RAROS, PUEDEN SER GRAVES

En 100 personas a quienes se les ha colocado una aguja intravenosa para la administración de un agente de contraste, 1 persona o menos pueden tener:

- Desvanecimiento (desmayo)
- Sangrado

#### Riesgos asociados con el agente de contraste o tinte radiográfico

#### OCASIONALES, PUEDEN SER GRAVES

En 100 personas que reciben un agente de contraste o tinte radiográfico, entre 4 y 20 personas pueden tener:

- Náuseas/vómitos
- Sensación de calidez o de rubefacción
- Erupción cutánea (sarpullido) o urticaria
- Picazón

#### RAROS, PUEDEN SER GRAVES

En 1000 personas que reciben un agente de contraste o tinte radiográfico, 1 persona o menos pueden tener:

Daño temporal en el riñón

#### MUY POCO FRECUENTES Y GRAVES

En 1,000,000 de personas que reciben un agente de contraste o tinte radiográfico, 4 personas menos pueden tener lo siguiente:

- Inflamación de la boca y la garganta
- Ritmo cardiaco anormal
- Desvanecimiento (desmayo) y presión arterial muy baja que requiere tratamiento

Puede haber otros efectos secundarios que los investigadores desconocen en este momento. Es importante que, si se detectan nuevos efectos secundarios, el médico del estudio los analice con usted.

Informe al médico del estudio sobre cualquier duda que tenga acerca de posibles efectos secundarios. Puede consultar al médico del estudio sobre los efectos secundarios en cualquier momento.

# ¿Cuáles son los posibles beneficios que puedo esperar de la participación en este estudio?

Este estudio de investigación solo tiene una pequeña posibilidad de ayudarla porque no sabemos si el examen de TAC de perfusión predice en forma precisa los efectos del bevacizumab. Este estudio de investigación puede ayudar a los investigadores a aprender cosas que podrían beneficiar a otras personas en el futuro.

## ¿Puedo dejar de participar en este estudio?

Sí. Puede decidir dejar de participar en cualquier momento. Si decide interrumpir la participación por cualquier motivo, es importante informar al médico del estudio tan pronto como sea posible para que pueda dejar de participar sin riesgos. Si deja de participar, puede decidir si desea, o no, que el médico del estudio siga brindando su información médica a la organización que está llevando a cabo el estudio.

El médico del estudio le notificará sobre información nueva o cambios en el estudio que pudieran afectar su salud o su deseo de continuar en el estudio.

El médico del estudio puede retirarla del estudio:

- Si se producen cambios en su salud y el estudio ya no es conveniente para usted
- Si surge información nueva
- Si usted no sigue las normas del estudio
- Si el patrocinador, el Consejo de revisión institucional o la Administración de Alimentos y Medicamentos (FDA, Food and Drug Administration) interrumpen el estudio.

### ¿Cuáles son mis derechos en este estudio?

La participación en este estudio de investigación es su elección. Independientemente de la decisión que tome, e incluso si cambia de decisión, no habrá penalidades para usted. No perderá su atención médica ni sus derechos legales.

#### ¿Cuáles son los costos de participar en este estudio?

No se le cobrarán las dos TAC de perfusión mientras participe en este estudio de investigación.

Usted o su plan de salud/compañía de seguro tendrá que pagar todos los demás costos del tratamiento de su cáncer mientras participa en este estudio de investigación; incluso el costo de la preparación y administración del fármaco del estudio, las pruebas, procedimientos o medicamentos para tratar los efectos secundarios, a menos que se le indique que determinadas pruebas se realizan sin costo. Antes de que decida participar en el estudio de investigación, debe consultar a su plan de salud o compañía de seguros para determinar con exactitud qué pagarán.

No se le pagará por participar en este estudio de investigación.

# ¿Qué sucede si me lesiono o sufro daños debido a mi participación en este estudio?

Si sufre lesiones o daño como consecuencia de su participación en este estudio de investigación y necesita tratamiento médico, informe al médico del estudio. Los patrocinadores del estudio no se ofrecerán a pagar por el tratamiento médico de las lesiones. Es posible que su compañía de seguros no esté dispuesta a pagar por una lesión relacionada con el estudio de investigación. Si no tiene seguro, usted será responsable de cualquier costo.

Si cree que esta lesión fue consecuencia de un error médico, usted conserva sus derechos legales de recibir el pago de esto incluso si está participando en un estudio de investigación.

## ¿Quién verá mi información médica?

Su privacidad es muy importante para nosotros y los investigadores harán todos los esfuerzos por protegerla. Si la ley lo exige, su información puede divulgarse. Por ejemplo, ciertos estados requieren que los médicos informen a las juntas médicas si detectan una enfermedad, como tuberculosis. Sin embargo, los investigadores harán todo lo posible para asegurarse de que cualquier información que se divulgue no la identifique. Parte de su información médica

o la información sobre su espécimen que se obtenga en este estudio se mantendrá en una base de datos central para la investigación. La base de datos no incluirá su nombre ni su información de contacto.

El grupo de investigación ECOG-ACRIN Cancer Research Group lleva a cabo este estudio. ECOG-ACRIN es un grupo de investigación del cáncer que realiza estudios para el Instituto Nacional del Cáncer. Su médico es miembro de ECOG-ACRIN u otro grupo que participa en este estudio. Para ayudar a proteger su privacidad, ECOG-ACRIN ha obtenido un Certificado de confidencialidad de parte del Departamento de Salud y Servicios Humanos (DHHS, Department of Health and Human Services). Con este Certificado, ECOG-ACRIN no puede verse obligado (por ejemplo, por medio de un citatorio judicial) a divulgar información que pudiera identificarla en ningún proceso federal, estatal o local de carácter civil, penal, administrativo, legislativo o de otro tipo. Sin embargo, la divulgación será necesaria ante la solicitud del DHHS para los fines de auditoría o evaluación del programa.

Existen organizaciones que pueden inspeccionar sus registros. Estas organizaciones están obligadas a garantizar que se mantenga la privacidad de su información, a menos que la ley les exija brindar información. Algunas de estas organizaciones son las siguientes:

- ECOG-ACRIN Cancer Research Group
- El Consejo de revisión institucional (CRI), un grupo de personas que revisa la investigación con el fin de proteger a las personas que participan en el estudio.
- La Administración de Alimentos y Medicamentos y el Instituto Nacional del Cáncer en los Estados Unidos, e instituciones similares si otros países participan del estudio.
- Harvard Tumor Imaging Metrics Core

### ¿Dónde puedo obtener más información?

Puede visitar el sitio web de NCI en <a href="http://cancer.gov/">http://cancer.gov/</a> para obtener más información sobre los estudios o información general sobre el cáncer. También puede llamar al servicio de información sobre cáncer del NCI para obtener la misma información en: 1-800-4-CANCER (1-800-422-6237).

Según lo exigen las leyes de los Estados Unidos, habrá una descripción de este ensayo clínico disponible en <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>. Este sitio web no incluirá información que pueda identificarla. Como máximo, el sitio web incluirá un resumen de los resultados. Puede hacer búsquedas en este sitio web en cualquier momento.

| ¿Quién puede res | sponder a mis preguntas sobre este estudio? |
|---|---|
| de este estudio o | el médico del estudio sobre cualquier pregunta o inquietud que tenga acerca para informar efectos secundarios o lesiones. Comuníquese con el médico (inserte el nombre del médico del estudio) al (inserte número de teléfono). |
| Mi firma para ac | eptar participar en el estudio principal |
| del estudio y se h | ha leído, este formulario de consentimiento. Lo he analizado con el médico an respondido mis preguntas. Se me entregará una copia firmada de este to participar en el estudio principal. |
| Firma de la partic | ipante |
| Fecha de la firma | |
| Firma de la perso | na que lleva a cabo la discusión del consentimiento informado |
| Fecha de la firma | |

# Título del estudio para los participantes del estudio: Evaluación de la TAC de perfusión para predecir la respuesta al tratamiento con bevacizumab en cáncer de ovarios, de trompas de Falopio y peritoneal

#### Título oficial del estudio para la búsqueda en Internet en

https://ClinicalTrials.gov: EAE161 Perfusion CT to Predict Progression-free Survival and Response Rate in Bevacizumab and Paclitaxel Treatment of Platinum-Resistant Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Carcinoma.

(EAE161 TAC de perfusión para predecir la supervivencia libre de progresión y la tasa de respuesta al tratamiento con bevacizumab y paclitaxel en carcinoma ovárico epitelial, de trompas de Falopio o peritoneal resistente a platino persistentes o recurrentes).

#### Consentimiento para la selección

Fecha de la versión: 13 de junio de 2018

# ¿Cuál es el enfoque habitual para el monitoreo de mi cáncer ovárico, de trompas de Falopio o peritoneal?

Se la invita a participar en este estudio de investigación porque están a punto de realizarle una tomografía computada (TAC) de tórax, abdomen y pelvis como parte de su atención de rutina. Las pruebas se realizan para determinar si su cáncer ovárico, de trompas de Falopio o peritoneal se puede observar a través de estudios de diagnóstico por imágenes. Si la TAC indica que tiene cáncer persistente o recurrente, su médico desea enviar las imágenes de TAC y la información sobre su tipo de tumor a los investigadores de ECOG-ACRIN Cancer Research Group, un grupo de investigación del Instituto Nacional del Cáncer. Los científicos de ECOG-ACRIN revisarán las imágenes de su TAC para determinar si usted reúne los requisitos para participar en un estudio de diagnóstico por imágenes ECOG-ACRIN. Si se determina que reúne los requisitos, su médico le explicará el estudio de diagnóstico por imágenes y, si decide participar en ese momento, se le pedirá que firme un formulario de consentimiento separado.

# ¿Cuáles son mis otras opciones si no participo en este estudio?

Si decide no participar en este estudio, tiene otras opciones para su atención. Por ejemplo:

- puede optar por recibir la atención habitual de rutina
- puede optar por participar en un estudio de investigación diferente, si hubiera uno disponible

#### ¿Por qué se realiza este estudio?

El objetivo de este formulario es obtener su permiso para determinar si es elegible para un ensayo. Le solicitamos su autorización para enviar imágenes de su TAC de tórax, abdomen y pelvis a ECOG-ACRIN. Se revisarán estas imágenes para determinar si es elegible para un ensayo de diagnóstico por imágenes donde se evaluará la TAC de perfusión, una prueba de diagnóstico por imágenes que observa el flujo de sangre al tumor. Mientras está en el equipo de tomografía, se le inyecta un agente de contraste en las venas y se obtienen muchas imágenes secuenciales de su tumor mientras el contraste fluye dentro y fuera del tumor. Para usted, la experiencia es similar a una TAC convencional, salvo que las imágenes que se obtienen en este estudio se concentran más en un área específica de su cuerpo, donde se ubica el tumor.

Si en esta prueba de detección se confirma que usted es elegible, el estudio de diagnóstico por imágenes se le explicará por separado. En ese momento, si decide participar en el estudio de diagnóstico por imágenes, se le pedirá que firme otro consentimiento. Si en esta prueba de detección se confirma que usted es no es elegible, ya no participará en este estudio. Recibirá tratamiento con la atención habitual.

Se seleccionará a aproximadamente 300 pacientes.

#### ¿Cuáles son los grupos del estudio?

Se realizará una TAC a todos los participantes del estudio de selección como parte de la atención habitual. Si en la TAC se observa que tiene cáncer recurrente o persistente, su TAC se utilizará para determinar si tiene una lesión que hace que sea elegible para un estudio de diagnóstico por imágenes para evaluar la TAC de perfusión. Estas imágenes se enviarán a ECOG-ACRIN donde se confirmará si es elegible para el estudio de diagnóstico por imágenes de ECOG-ACRIN.

Lea el cuadro a continuación como otra manera de conocer qué le pasará durante este estudio de investigación. Empiece a leer de izquierda a derecha, siguiendo las líneas y flechas.

#### Selección



### ¿Durante cuánto tiempo participaré en este estudio?

Una vez que se envíen las imágenes de la TAC a ECOG-ACRIN, el grupo de investigación revisará las imágenes en un plazo de cinco días hábiles. ECOG-ACRIN le informará a su médico si es elegible para el estudio de diagnóstico por imágenes de TAC de perfusión. Si es elegible, se llevará a cabo una discusión y un proceso de consentimiento separados. Si se determina que es elegible y se inscribe en el estudio, la participación en este se extenderá por un mínimo de 18 meses y un máximo de tres años y medio.

# ¿Qué pruebas y procedimientos adicionales se me realizarán si participo en este estudio?

Será necesario realizarle un análisis de sangre para revisar la función renal. Las pruebas que se le realizan forman parte de la atención habitual para su cáncer.

# ¿Cuáles son los posibles riesgos que puedo esperar de la participación en este estudio?

Si decide participar en este estudio de investigación, existe el riesgo de lo siguiente:

- Su información médica se divulgue o utilice erróneamente. Este es un riesgo pequeño, ya que su información médica está protegida, pero sigue existiendo el riesgo.
- Pueda perder tiempo de trabajo o en su hogar y pasar más tiempo en el hospital o en el consultorio médico de lo habitual.
- Si la TAC muestra un tumor, su tratamiento puede demorarse hasta cinco días mientras se aguardan los resultados de esta selección.

# ¿Cuáles son los posibles beneficios que puedo esperar de la participación en este estudio?

No se espera que esta selección la beneficie.

## ¿Puedo dejar de participar en este estudio?

Sí. Puede decidir dejar de participar en cualquier momento. Si decide interrumpir la participación por cualquier motivo, es importante informar al médico del estudio tan pronto como sea posible para que pueda dejar de participar sin riesgos. Si deja de participar, puede decidir si desea, o no, que el médico del estudio siga brindando su información médica a la organización que está llevando a cabo el estudio.

El médico del estudio le notificará sobre información nueva o cambios en el estudio que pudieran afectar su salud o su deseo de continuar en el estudio.

El médico del estudio puede retirarla del estudio:

- Si surge información nueva
- Si usted no sigue las normas del estudio
- Si el patrocinador, el Consejo de revisión institucional o la Administración de Alimentos y Medicamentos (FDA, Food and Drug Administration) interrumpen el estudio.

#### ¿Cuáles son mis derechos en este estudio?

La participación en este estudio de investigación es su elección. Independientemente de la decisión que tome, e incluso si cambia de decisión, no habrá penalidades para usted. No perderá su atención médica ni sus derechos legales.

| Si tiene preguntas sobre su | s derechos mientras participa en | este estudio, llame al Consejo |
|---|---|---|
| de revisión institucional de | | (insert name of center) |
| al | <mark>(insert telephone number</mark> ). (Note | to Local Investigator: Contact |
| information for patient rep | resentatives or other individuals | at a local institution who are not |
| on the IRB or research tear | n but take calls regarding clinica | l trial questions can also be listed |
| here.) | | |

#### ¿Cuáles son los costos de participar en este estudio?

Usted o su plan de salud/compañía de seguro tendrá que pagar todos los demás costos del tratamiento de su cáncer mientras participa en este estudio de investigación; incluso el costo de la preparación y administración del fármaco del estudio, las pruebas, procedimientos o medicamentos para tratar los efectos secundarios, a menos que se le indique que determinadas pruebas se realizan sin costo. Antes de que decida participar en el estudio de investigación, debe consultar a su plan de salud o compañía de seguros para determinar con exactitud qué pagarán.

No se le pagará por participar en este estudio de investigación de selección. La revisión de su TAC por parte de ECOG-ACRIN se llevará a cabo sin costo para usted ni para su seguro. No será responsable del costo del examen de TAC de perfusión, el examen de función renal ni los análisis de sangre para evaluar los niveles de CA-125.

# ¿Qué sucede si me lesiono o sufro daños debido a mi participación en este estudio?

Si sufre lesiones o daño como consecuencia de su participación en este estudio de investigación y necesita tratamiento médico, informe al médico del estudio. Los patrocinadores del estudio no se ofrecerán a pagar por el tratamiento médico de las lesiones. Es posible que su compañía de seguros no esté dispuesta a pagar por una lesión relacionada con el estudio de investigación. Si no tiene seguro, usted será responsable de cualquier costo.

Si cree que esta lesión fue consecuencia de un error médico, usted conserva sus derechos legales de recibir el pago de esto incluso si está participando en un estudio de investigación.

#### ¿Quién verá mi información médica?

Su privacidad es muy importante para nosotros y los investigadores harán todos los esfuerzos por protegerla. Si la ley lo exige, su información puede divulgarse. Por ejemplo, ciertos estados requieren que los médicos informen a las juntas médicas si detectan una enfermedad, como tuberculosis. Sin embargo, los investigadores harán todo lo posible para asegurarse de que cualquier información que se divulgue no la identifique. Parte de su información médica o la información sobre su espécimen que se obtenga en este estudio se mantendrá en una base de datos central para la investigación. La base de datos no incluirá su nombre ni su información de contacto.

El grupo de investigación ECOG-ACRIN Cancer Research Group lleva a cabo este estudio. ECOG-ACRIN es un grupo de investigación del cáncer que realiza estudios para el Instituto Nacional del Cáncer. Su médico es miembro de ECOG-ACRIN u otro grupo que participa en este estudio. Para ayudar a proteger su privacidad, ECOG-ACRIN ha obtenido un Certificado de confidencialidad de parte del Departamento de Salud y Servicios Humanos (DHHS, Department of Health and Human Services). Con este Certificado, ECOG-ACRIN no puede verse obligado (por ejemplo, por medio de un citatorio judicial) a divulgar información que pudiera identificarla en ningún proceso federal, estatal o local de carácter civil, penal, administrativo, legislativo o de otro tipo. Sin embargo, la divulgación será necesaria ante la solicitud del DHHS para los fines de auditoría o evaluación del programa.

Existen organizaciones que pueden inspeccionar sus registros. Estas organizaciones están obligadas a garantizar que se mantenga la privacidad de su información, a menos que la ley les exija brindar información. Algunas de estas organizaciones son las siguientes:

- El Consejo de revisión institucional (CRI), un grupo de personas que revisa la investigación con el fin de proteger a las personas que participan en el estudio.
- La Administración de Alimentos y Medicamentos y el Instituto Nacional del Cáncer en los Estados Unidos, e instituciones similares si otros países participan del estudio.
- Harvard Tumor Metrics Imaging Core
- ECOG-ACRIN Cancer Research Group

### ¿Dónde puedo obtener más información?

Puede visitar el sitio web de NCI en <a href="http://cancer.gov/">http://cancer.gov/</a> para obtener más información sobre los estudios o información general sobre el cáncer. También puede llamar al Servicio de información sobre cáncer del NCI para obtener la misma información en: 1-800-4-CANCER (1-800-422-6237).

Según lo exigen las leyes de los Estados Unidos, habrá una descripción de este ensayo clínico disponible en <a href="https://ClinicalTrials.gov">https://ClinicalTrials.gov</a>. Este sitio web no incluirá información que pueda identificarla. Como máximo, el sitio web incluirá un resumen de los resultados. Puede hacer búsquedas en este sitio web en cualquier momento.

| der a mis preguntas sobre este estudio? |
|---|
| édico del estudio sobre cualquier pregunta o inquietud que tenga acerca nformar efectos secundarios o lesiones. Comuníquese con el médico (insert name of study doctor[s]) al insert telephone number). |
| r participar en el estudio |
| rído, este formulario de consentimiento. Lo he analizado con el médico spondido mis preguntas. Se me entregará una copia firmada de este ticipar en la porción de selección de este estudio. |
| e |
| e lleva a cabo la discusión del consentimiento informado |
| i i i i i i i i i i i i i i i i i i i |